CLINICAL TRIAL: NCT01872689
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Study to Assess the Efficacy and Safety of Lebrikizumab in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Study of Lebrikizumab in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB28547; 2013-001163-24 (EudraCT Number)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — lebrikizumab; pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Monotherapy (Cohort A): Placebo (Placebo Comparator): Participants will receive monotherapy with placebo matched to lebrikizumab administered via subcutaneous (SC) injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period. Participants will be allowed to receive treatment with lebrikizumab at a dose of 250 mg administered via SC injection once every 4 weeks up to additional 52 weeks (that is, up to Week 104) in the open-label period.
  Interventions: Drug: Lebrikizumab; Drug: Placebo
- Monotherapy (Cohort A): Lebrikizumab (Experimental): Participants will receive monotherapy with lebrikizumab at a dose of 250 milligrams (mg) administered via SC injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period. Participants will be allowed to receive treatment with lebrikizumab at a dose of 250 mg administered via SC injection once every 4 weeks up to additional 52 weeks (that is, up to Week 104) in the open-label period.
  Interventions: Drug: Lebrikizumab
- Combination Therapy (Cohort B): Placebo + Pirfenidone (Placebo Comparator): Participants will receive pirfenidone at a stable dose of 2403 mg per day (three 267 mg capsules three times a day [9 capsules daily] for a total of 2403 mg/day) or at maximum tolerated dose (MTD) administered orally along with placebo matched to lebrikizumab administered via SC injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period.
  Interventions: Drug: Pirfenidone; Drug: Placebo
- Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone (Experimental): Participants will receive pirfenidone at a stable dose of 2403 mg per day (three 267 mg capsules three times a day [9 capsules daily] for a total of 2403 mg/day) or at MTD administered orally along with lebrikizumab at a dose of 250 mg administered via SC injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period.
  Interventions: Drug: Lebrikizumab; Drug: Pirfenidone

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab will be administered at a dose of 250 mg via SC injection once every 4 weeks.
  Other Names: RO5490255
  Arms: Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; Monotherapy (Cohort A): Lebrikizumab; Monotherapy (Cohort A): Placebo
Drug: Pirfenidone — Pirfenidone will be administered orally at a stable dose of 2403 mg per day or at MTD.
  Arms: Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; Combination Therapy (Cohort B): Placebo + Pirfenidone
Drug: Placebo — Placebo matched to lebrikizumab will be administered via SC injection once every 4 weeks.
  Arms: Combination Therapy (Cohort B): Placebo + Pirfenidone; Monotherapy (Cohort A): Placebo

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy and safety of lebrikizumab as monotherapy in the absence of background IPF therapy and as combination therapy with pirfenidone background therapy in participants with IPF. Participants will be randomized to receive either lebrikizumab or placebo subcutaneously every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of IPF within the previous 5 years from time of screening and confirmed at baseline
* FVC >/=40 percent (%) and </=100% of predicted at screening
* Stable baseline lung function as evidenced by a difference of less than (<) 10% in FVC (in liters) measurements between screening and Day 1, Visit 2 prior to randomization
* DLco >/=25% and </=90% of predicted at screening
* Ability to walk >/=100 meters unassisted in 6 minutes
* Cohort A: No background IPF therapy for >/=4 weeks allowed prior to randomization and throughout the placebo-controlled study period
* Cohort B: Tolerated dose of pirfenidone </=2403 milligrams once daily (mg/day) for >/=4 weeks required prior to randomization and throughout the placebo-controlled study period

Exclusion Criteria:

* History of severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Evidence of other known causes of interstitial lung disease
* Lung transplant expected within 12 months of screening
* Evidence of clinically significant lung disease other than IPF
* Post-bronchodilator forced expiratory volume in 1 second (FEV1)/FVC ratio <0.7 at screening
* Positive bronchodilator response, evidenced by an increase of >/=12% predicted and 200 milliliters increase in FEV1 or FVC
* Class IV New York Heart Association chronic heart failure or historical evidence of left ventricular ejection fraction <35%
* Hospitalization due to an exacerbation of IPF within 4 weeks prior to or during screening
* Known current malignancy or current evaluation for potential malignancy
* Listeria monocytogenes infection or active parasitic infection within 6 months prior to Day 1, Visit 2
* Active tuberculosis requiring treatment within 12 months of screening
* Known immunodeficiency, including but not limited to human immunodeficiency virus infection
* Past use of any anti-interleukin (IL)-13 or anti-IL-4/IL-13 therapy, including lebrikizumab
* Evidence of acute or chronic hepatitis or known liver cirrhosis

Exclusions Criteria Limited to Cohort B:

* Known achalasia, esophageal stricture, or esophageal dysfunction sufficient to limit the ability to swallow oral medication
* Tobacco smoking or use of tobacco-related products within 3 months of screening or unwillingness to avoid smoking throughout the study period
* Known or suspected peptic ulcer
* Any condition that, as assessed by the investigator, might be significantly exacerbated by the known side effects associated with pirfenidone
* Creatinine clearance <40 milliliters/minute, calculated using the Cockcroft-Gault formula
* Use of following therapies within 4 weeks of randomization (Day 1, Visit 2) or during the study: Strong inhibitors of CYP1A2 (Cytochrome P450 Family 1 Subfamily A Member 2) (example: fluvoxamine or enoxacin); Moderate inducers of CYP1A2 (limited to tobacco smoking and tobacco-related products)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2013-10-13 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (112):
- United States (54):
  - University Alabama At Birmingham, Birmingham, Alabama
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - Southern Arizona Veterans Administration Healthcare Systems, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - UCSD Medical Center, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Rocky Mountain Center For Clinical Research, Wheat Ridge, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Research Alliance Inc, Clearwater, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - University Miami, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - USF Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Healthcare Pulmonary and Critical Care Research, Austell, Georgia
  - Southeastern Lung Care, Decatur, Georgia
  - University of Chicago; Pulmonary and Critical Care, Chicago, Illinois
  - Loyola University Med Center, Maywood, Illinois
  - Univ of Iowa Hosp & Clinics; Pulmonary, Iowa City, Iowa
  - Uni of Kansas Medical Center, Kansas City, Kansas
  - Via Christi Hospital Inc. DBA Via Christi Research; Research Dept., Wichita, Kansas
  - Maine Medical Center -Division of Pulmomary and Critical Care Medicine, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center - Johns Hopkins Asthma & Allergy Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota Hospital & Clinic, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Cardiopulmonary Associates LLC Cardiopulmonary Research, Chesterfield, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Weill Medical College of Cornell University, New York, New York
  - Mt Sinai School Medical Pulmo And Critical Care Med, New York, New York
  - Highland Hospital-University of Rochester Medical Center, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Research University; University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - The Oregon Clinic., Portland, Oregon
  - Penn State University College Medical Allergy And Care Med, Hershey, Pennsylvania
  - Temple Lung Center, Temple Universtiy-Of the Commomwealth System of Higher Education, Philadelphia, Pennsylvania
  - University of Pittsburgh Med Cen; Dorothy P And Richard P Simmons Cen For Interstitial Lung Disease, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College Med, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Audie Murphy Va Hospital, San Antonio, Texas
  - University of Utah Health Sciences Center, Lung Health Research Center, Salt Lake City, Utah
  - University Vermont College Medicine Fletcher Allen Health Care, Colchester, Vermont
  - Inova Transplant Center Fairfax Hospital, Falls Church, Virginia
  - Pulmonary Consultants, Tacoma, Washington
  - University Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Royal Prince Alfred Hospital; Department of Respiratory Medicine, Camperdown, New South Wales
  - ST VINCENT'S HOSPITAL; Thoracic Medicine, Darlinghurst, New South Wales
  - Box Hill Hospital; Eastern Clinical Research Unit, Box Hill, Victoria
  - Alfred Hospital; Allergy Immuno Resp, Melbourne, Victoria
  - Institute for Respiratory Health Inc, Nedlands, Western Australia
- Belgium (4):
  - Hospital Erasme; Neurologie, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - CHU UCL Mont-Godinne, Mont-godinne
- Canada (5):
  - University of British Columbia - Vancouver Coastal Health Authority, Vancouver, British Columbia
  - Dr. Georges-L. Dumont Regional Hospital, Moncton, New Brunswick
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Lawson Health Research Institute a joint venture of LHSC Research Inc and Lawson Research Institute, London, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec (Hôpital Laval), Ste. Foy, Quebec
- France (5):
  - Hopital Avicenne; Pneumologie, Bobigny
  - Hopital Louis Pradel; Pneumologie, Bron
  - Hopital Calmette; Pneumologie, Lille
  - Hopital Bichat Claude Bernard ; Service de Pneumologie, Paris
  - Hopital de Pontchaillou; Service de Pneumologie, Rennes
- Germany (6):
  - Ruhrlandklinik Lungenzentrum der UNI Essen Abt.Pneumologie-Allergologie, Essen
  - Universitätsklinikum Standort Gießen Medizinische Klinik II u. Poliklinik Innere Med./Pneumologie, Giessen
  - LungenClinic Großhansdorf, Großhansdorf
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - CPC Comprehensive Pneumology Center / Forschungsambulanz, Helmholtz Zentrum, München
- Italy (6):
  - Ospedale Morgagni-Pierantoni; U.O. Pneumologia, Forlì, Emilia-Romagna
  - Policlinico Tor Vergata; UO Mal. Respiratorie; Centro Malattie rare polmone, Rome, Lazio
  - Ospedale San Giuseppe; U.O. di Pneumologia, Milan, Lombardy
  - A.O. Universitaria San Luigi Gonzaga di Orbassano; Ambulatorio per le Malattie Rare del Polmone, Orbassano (TO), Piedmont
  - A.O.U. Policlinico Vittorio Emanuele; Centro per la cura delle Malattie Rare del Polmone, Catania, Sicily
  - A.O. Univ. Senese Policlinico S. Maria alle Scotte; UOC Malattie Resepiratorie e Trapianto Polmonare, Siena, Tuscany
- Japan (3):
  - Kanagawa Cardiovascular and Respiratory Center; Respiratory Medicine, Kanagawa
  - Kinki-Chuo Chest Medical Center, Osaka
  - Tosei General Hospital, Seto-shi
- Mexico (4):
  - Hospital General Del Estado De Sonora "Dr. Ernesto Ramos Bours"; Servicio De Neumologia, Hermosillo
  - Instituto Nacional De Enfermedades Respiratorias;Unidad de Investigación, Mexico City
  - Universidad Autonoma De Nuevo Leon, Hospital Universitario Doctor Jose Eleuterio Gonzalez, Monterrey
  - Unidad de Investigacion Clinica En Medicina (Udicem) S.C., Monterrey
- Peru (3):
  - Clinica San Pablo, Lima
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
  - Clinica San Borja; NEUMOCARE, Lima
- Poland (5):
  - Uniwersytecki Szpital Kliniczny Nr 1 im.N.Barlickiego Oddzial Kliniczny Pneumonologii i Alergologii, Lodz
  - Ms Clinsearch Specjalistyczny Niepubliczny Zaklad Opieki Zdrowotnej, Lublin
  - Klinika Pulmonologii, Alergologii i Onkologii Pulmonologicznej Uniwersytet Medyczny w Poznaniu, Poznan
  - Instytut Gruzlicy i Chorob Płuc, Warsaw
  - Klinika Chorob Pluc i Gruzlicy w Zabrzu; Slaski Uniwersytet Medyczny, Zabrze
- Spain (5):
  - Hospital Universitari de Bellvitge ; Servicio de Neumologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario La Princesa; Servicio de Neumologia, Madrid
  - Hospital Clínico San Carlos - Servicio de Neumologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Neumologia, Seville
  - Hospital General Universitario De Valencia; Servicio de Neumologia, Valencia
- United Kingdom (7):
  - Southmead Hospital; Respiratory Department, Bristol
  - Papworth Hospital NHS Foundation Trust; Respiratory Department, Cambridge
  - Southampton General Hospital; Respiratory Department, Hampshire
  - St James University Hospital; Respiratory Department, Leeds
  - Respiratory research department clinical science building, Liverpool
  - Royal Brompton Hospital; Respiratory Department, London
  - North Manchester Hospital; Respiratory Department, Manchester

REFERENCES:
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 505 participants (154 participants in Monotherapy Cohort and 351 participants in Combination Therapy Cohort) were enrolled in the study.
Groups:
- Monotherapy (Cohort A): Placebo: Participants received monotherapy with placebo matched to lebrikizumab administered via subcutaneous (SC) injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period. Participants were allowed to receive treatment with lebrikizumab at a dose of 250 milligrams (mg) administered via SC injection once every 4 weeks up to additional 52 weeks (that is, up to Week 104) in the open-label period.
- Monotherapy (Cohort A): Lebrikizumab: Participants received monotherapy with lebrikizumab at a dose of 250 mg administered via SC injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period. Participants were allowed to receive treatment with lebrikizumab at a dose of 250 mg administered via SC injection once every 4 weeks up to additional 52 weeks (that is, up to Week 104) in the open-label period.
- Combination Therapy (Cohort B): Placebo + Pirfenidone: Participants received pirfenidone at a stable dose of 2403 mg per day (three 267 mg capsules three times a day [9 capsules daily] for a total of 2403 mg/day) or at maximum tolerated dose (MTD) administered orally along with placebo matched to lebrikizumab administered via SC injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period.
- Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone: Participants received pirfenidone at a stable dose of 2403 mg per day (three 267 mg capsules three times a day [9 capsules daily] for a total of 2403 mg/day) or at MTD administered orally along with lebrikizumab at a dose of 250 mg administered via SC injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period.
Period: Double-Blind/Placebo-Controlled Period
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Started | 76 | 78 | 177 | 174
Completed | 56 | 58 | 129 | 136
Not Completed | 20 | 20 | 48 | 38
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 6 | 3
Not completed — Withdrawal by Subject | 9 | 8 | 14 | 16
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 3 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Death | 3 | 4 | 14 | 9
Not completed — Adverse Event | 6 | 3 | 10 | 7
Period: Open-Label Period (Only For Monotherapy)
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Started | 52 (Of the 56 participants who completed Period 1, only 52 started Period 2.) | 56 (Of the 58 participants who completed Period 1, only 56 started Period 2.) | 0 (As per study design, Period 2 was not intended for this arm.) | 0 (As per study design, Period 2 was not intended for this arm.)
Completed | 31 | 33 | 0 | 0
Not Completed | 21 | 23 | 0 | 0
Not completed — Other | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 12 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0
Not completed — Death | 5 | 3 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-Treat (ITT) Population, which included all participants who were randomized in the study, with participants grouped according to the treatment assignment at randomization.
Groups:
- Monotherapy (Cohort A): Placebo: Participants received monotherapy with placebo matched to lebrikizumab administered via SC injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period. Participants were allowed to receive treatment with lebrikizumab at a dose of 250 mg administered via SC injection once every 4 weeks up to additional 52 weeks (that is, up to Week 104) in the open-label period.
- Combination Therapy (Cohort B): Placebo + Pirfenidone: Participants received pirfenidone at a stable dose of 2403 mg per day (three 267 mg capsules three times a day [9 capsules daily] for a total of 2403 mg/day) or at MTD administered orally along with placebo matched to lebrikizumab administered via SC injection once every 4 weeks up to 52 weeks during the placebo-controlled treatment period.
- Total: Total of all reporting groups
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone | Total
Number analyzed (Participants) | 76 | 78 | 177 | 174 | 505
Age, Customized [Number; unit: participants]
  From 40 to <55 years | 2 | 1 | 6 | 2 | 11
  From 55 to <65 years | 18 | 10 | 40 | 41 | 109
  From 65 to <75 years | 38 | 44 | 99 | 92 | 273
  >/=75 years | 18 | 23 | 32 | 39 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 30 | 37 | 93
  Male | 63 | 65 | 147 | 137 | 412
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 13 | 15 | 43
  Not Hispanic or Latino | 64 | 68 | 160 | 155 | 447
  Unknown or Not Reported | 3 | 4 | 4 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 1 | 3
  Asian | 11 | 8 | 19 | 15 | 53
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 60 | 66 | 149 | 151 | 426
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 3 | 2 | 7 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Decrease in Percent Predicted Forced Vital Capacity (FVC) Over 52 Weeks
Description: Annualized rates of decrease (slope throughout time from baseline to Week 52) for percent predicted FVC was assessed and reported. FVC is a standard pulmonary function test. FVC is defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted FVC is based on sex, age, and height of a person. Percent predicted FVC (in %) = [(observed FVC)/(predicted FVC)]*100.
Time Frame: Baseline up to Week 52 (assessed at Baseline, Weeks 1, 4, 12, 24, 36, 44, and 52)
Population: Analysis was performed on ITT Population. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure at Week 52.
Measure: Mean (Standard Error); unit: percent predicted FVC/year
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 53 | 56 | 120 | 134
percent predicted FVC/year | -6.1876 (0.92597) | -5.2065 (0.92758) | -6.0430 (0.60633) | -5.5430 (0.59507)
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; Mixed Linear model comparing Lebrikizumab to Placebo, with assessment as the outcome variable; assessment time by treatment as fixed effects; and participant baseline FVC (<50%, 50 to 75%, >75%) and participant by assessment time as random effects with unstructured covariance; Test type: Superiority; p = 0.4555, Mixed Models Analysis; Median Difference (Final Values) = 0.98111, 95% CI 2-sided [-1.61 to 3.57], Standard Error of Mean 1.31064
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5566, Mixed Models Analysis; Mean Difference (Final Values) = 0.49998, 95% CI 2-sided [-1.17 to 2.17], Standard Error of Mean 0.84946

2. Secondary Outcome: Annualized Rate of Decline in 6-Minute Walk Test (6MWT) Distance Over 52 Weeks
Description: Annualized rates of decline (slope throughout time from baseline to Week 52) in 6MWT was assessed and reported. 6MWT was the distance (in meters [m]) that a participant could walk in 6 minutes.
Time Frame: Baseline up to Week 52 (assessed at Baseline, Weeks 1, 4, 12, 24, 36, 44, and 52)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: m/year
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 52 | 59 | 120 | 129
m/year | -44.6512 (15.97862) | -22.7209 (15.34753) | -25.5683 (12.24923) | -46.9810 (11.84199)
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3129, Mixed Models Analysis; Median Difference (Final Values) = 21.93023, 95% CI 2-sided [-20.97 to 64.83], Standard Error of Mean 21.62248
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2036, Mixed Models Analysis; Mean Difference (Final Values) = -21.4127, 95% CI 2-sided [-54.50 to 11.67], Standard Error of Mean 16.80160

3. Secondary Outcome: Percentage of Participants With Event of Greater Than or Equal to (>/=) 10% Absolute Decline in Percent Predicted FVC or Death From Any Cause
Description: FVC is defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted FVC is based on sex, age, and height of a person. Percent predicted FVC (in %) = [(observed FVC)/(predicted FVC)]*100.
Time Frame: Baseline up to the event of >/=10% absolute decline in percent predicted FVC or death from any cause, whichever occurred first (up to Week 122)
Population: Analysis was performed on ITT Population. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 76 | 76 | 175 | 173
percentage of participants | 34.2 | 27.6 | 30.3 | 26.6

4. Secondary Outcome: Time to First Occurrence of a >/=10% Absolute Decline in Percent Predicted FVC or Death From Any Cause
Description: FVC is defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted FVC is based on sex, age, and height of a person. Percent predicted FVC (in %) = [(observed FVC)/(predicted FVC)]*100. Time from randomization to first occurrence of an event of >/=10% absolute decline in percent predicted FVC or death from any cause was reported. Participants without an event were censored at the last assessment during the double-blind treatment period. Any participant who underwent lung transplantation was censored at the date of the transplant. The median time to event was estimated using Kaplan-Meier method. 95% confidence interval (CI) for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 76 | 76 | 175 | 173
weeks | 53.1 [52.6 to NA] — Upper limit of 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [52.9 to NA] — Median and upper limit of 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants.
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.4299, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.44 to 1.41]
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.3751, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.56 to 1.24]

5. Secondary Outcome: Annualized Rate of Decrease in Diffusion Capacity of the Lung for Carbon Monoxide (DLco) Over 52 Weeks
Description: Annualized rates of decrease (slope throughout time from baseline to Week 52) in DLco was assessed and reported. DLco (in milliliters per minute/millimeters of mercury [mL/min/mmHg]) is a measure of the gas transfer.
Time Frame: Baseline up to Week 52 (assessed at Baseline, Weeks 1, 4, 12, 24, 36, 44, and 52)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mL/min/mmHg/year
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 50 | 52 | 112 | 122
mL/min/mmHg/year | -4.7818 (0.74479) | -4.2400 (0.73826) | -5.7552 (0.46561) | -5.5732 (0.45577)
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6075, Mixed Models Analysis; Median Difference (Final Values) = 0.54171, 95% CI 2-sided [-1.54 to 2.62], Standard Error of Mean 1.05201
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7803, Mixed Models Analysis; Mean Difference (Final Values) = 0.18203, 95% CI 2-sided [-1.10 to 1.47], Standard Error of Mean 0.65206

6. Secondary Outcome: Percentage of Participants With Event of Death, All Cause Hospitalization, or a Decrease From Baseline of >/=10% in FVC
Description: FVC is defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted FVC is based on sex, age, and height of a person. Percent predicted FVC = [(observed FVC)/(predicted FVC)]*100.
Time Frame: Baseline up to the event of death from any cause, all cause hospitalization, or a decrease from baseline of >/=10% in FVC, whichever occurred first (up to Week 122)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 76 | 76 | 175 | 173
percentage of participants | 47.4 | 32.9 | 39.4 | 39.9

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: FVC is defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted FVC is based on sex, age, and height of a person. Percent predicted FVC = [(observed FVC)/(predicted FVC)]*100. PFS was defined as time from randomization to death from any cause, all cause hospitalization, or a decrease from baseline of >/=10% in FVC, whichever occurred first. Participants without an event were censored at the last assessment during the double-blind treatment period. Any participant who underwent lung transplantation was censored at the date of the transplant. The median PFS was estimated using Kaplan-Meier method. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 76 | 76 | 175 | 173
weeks | 52.6 [43.9 to NA] — Upper limit of 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [52.3 to NA] — Median and upper limit of 95% CI could not be estimated due to high number of censored participants.
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.0972, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.39 to 1.09]
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.9344, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.72 to 1.42]

8. Secondary Outcome: Annualized Rate of Decrease in FVC Over 52 Weeks
Description: Annualized rates of decrease (slope throughout time from baseline to Week 52) in FVC (in milliliters per year [mL/year]) was assessed and reported. FVC is defined as the volume of air that can forcibly be blown out after full inspiration in the upright position.
Time Frame: Baseline up to Week 52 (assessed at Baseline, Weeks 1, 4, 12, 24, 36, 44, and 52)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mL/year
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 53 | 57 | 120 | 134
mL/year | -221.029 (34.87511) | -192.906 (34.93853) | -231.167 (22.67786) | -209.437 (22.25073)
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5707, Mixed Models Analysis; Median Difference (Final Values) = 28.12302, 95% CI 2-sided [-69.80 to 126.04], Standard Error of Mean 49.47253 — Mean Difference = Lebrikizumab - Placebo
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4934, Mixed Models Analysis; Mean Difference (Final Values) = 21.72972, 95% CI 2-sided [-40.65 to 84.11], Standard Error of Mean 31.68767 — Mean Difference = Lebrikizumab - Placebo

9. Secondary Outcome: Annualized Rate of Decrease in A Tool to Assess Quality of Life in IPF (ATAQ-IPF) Questionnaire Total Score Over 52 Weeks
Description: The ATAQ-IPF Version 3 was utilized that included 31 items within 5 domains: cough (6 items), dyspnea (7 items), exhaustion (6 items), emotional well-being (6 items), and independence (6 items). Each item was assessed on a scale ranging from 1 (Strongly disagree) to 4 (Strongly agree). The ATAQ-IPF had a recall specification of 2 weeks. Simple summation scoring was used to derive individual domain scores as well as a total score. ATAQ-IPF total score ranged from 31 to 124 with lower score indicating better quality of life (QoL). Annualized rates of decrease (slope throughout time from baseline to Week 52) in ATAQ-IPF questionnaire total score was assessed and reported.
Time Frame: Baseline up to Week 52 (assessed at Baseline, Weeks 1, 4, 12, 24, 36, 44, and 52)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale/year
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 58 | 62 | 136 | 144
units on a scale/year | 6.8907 (1.71778) | 4.7886 (1.70370) | 5.6189 (0.99880) | 5.4558 (0.97793)
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3854, Mixed Models Analysis; Median Difference (Final Values) = -2.10204, 95% CI 2-sided [-6.88 to 2.68], Standard Error of Mean 2.41325
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9057, Mixed Models Analysis; Mean Difference (Final Values) = -0.16313, 95% CI 2-sided [-2.87 to 2.55], Standard Error of Mean 1.37698

10. Secondary Outcome: Percentage of Participants With an Event of St. George's Respiratory Questionnaire (SGRQ) Total Score Worsening or Death From Any Cause
Description: The SGRQ is a 50-item health-related QoL instrument that measured health impairment. The questionnaire contains 3 domains: symptoms, activity, and impacts. Items were assessed on various response scales, including a 5-point Likert scale and True/False scale. The SGRQ had a recall specification of 4 weeks. The SGRQ total score (summed weights) ranged from 0 to 100 with a lower score denoting a better health status. Percentage of participants with an event of SGRQ total score worsening (defined as reaching minimal important difference [MID], that is, an increase in total score of >/=7) or death from any cause was reported.
Time Frame: Baseline up to the event of SGRQ total score worsening or death from any cause, whichever occurred first (up to Week 122)
Population: Analysis was performed on ITT Population for monotherapy cohort only. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab
Number analyzed (Participants) | 76 | 76
percentage of participants | 57.9 | 48.7

11. Secondary Outcome: Time to First Occurrence of SGRQ Total Score Worsening or Death From Any Cause
Description: The SGRQ is a 50-item health-related QoL instrument that measured health impairment. The questionnaire contains 3 domains: symptoms, activity, and impacts. Items were assessed on various response scales, including a 5-point Likert scale and True/False scale. The SGRQ had a recall specification of 4 weeks. The SGRQ total score (summed weights) ranged from 0 to 100 with a lower score denoting a better health status. Time from randomization to first occurrence of an event of SGRQ total score worsening (defined as reaching minimal important difference [MID], that is, an increase in total score of >/=7) or death from any cause was reported. The median time to event was estimated using Kaplan-Meier method. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab
Number analyzed (Participants) | 76 | 76
weeks | 51.7 [24.1 to 54.6] | 52.3 [35.7 to NA] — Upper limit of 95% CI could not be estimated due to high number of censored participants.
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.4433, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.54 to 1.31]

12. Secondary Outcome: Percentage of Participants With an Event of Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbation
Description: IPF exacerbation was defined as an event that met all of the following criteria as determined by the investigator: Unexplained worsening or development of dyspnea within the previous 30 days; And radiologic evidence of new bilateral ground-glass abnormality or consolidation, superimposed on a reticular or honeycomb background pattern, that is consistent with usual interstitial pneumonitis; And absence of alternative causes, such as left heart failure, pulmonary embolism, pulmonary infection (on the basis of endotracheal aspirate or bronchoalveolar lavage if available, or investigator judgment), or other events leading to acute lung injury (for example, sepsis, aspiration, trauma, reperfusion pulmonary edema).
Time Frame: Baseline up to the event of acute IPF exacerbation (up to Week 122)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 76 | 76 | 175 | 172
percentage of participants | 3.9 | 3.9 | 6.3 | 2.9

13. Secondary Outcome: Time to First Event of Acute IPF Exacerbation
Description: Time from randomization to first occurrence of an event of IPF exacerbation was reported. IPF exacerbation was defined as an event that met all of the following criteria as determined by the investigator: Unexplained worsening or development of dyspnea within the previous 30 days; And radiologic evidence of new bilateral ground-glass abnormality or consolidation, superimposed on a reticular or honeycomb background pattern, that is consistent with usual interstitial pneumonitis; And absence of alternative causes, or other events leading to acute lung injury. The median time to event was estimated using Kaplan-Meier method. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Baseline up to the event of acute IPF exacerbation (up to Week 122)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 76 | 76 | 175 | 172
weeks | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants.
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.9366, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.21 to 5.30]
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.1346, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.16 to 1.31]

14. Secondary Outcome: Percentage of Participants With Respiratory-Related Hospitalization
Time Frame: Baseline up to the event of respiratory-related hospitalization (up to Week 122)
Population: Analysis was performed on ITT Population for combination therapy cohorts only. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 175 | 173
percentage of participants | 15.4 | 14.5

15. Secondary Outcome: Time to Respiratory-Related Hospitalization
Description: Time from randomization to first occurrence of an event of respiratory-related hospitalization was reported. Participants without an event were censored at the last known alive day, study Day 368, or the last date during the double-blind period. The median time to event was estimated using Kaplan-Meier method. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Baseline up to the event of respiratory-related hospitalization (up to Week 122)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 175 | 173
weeks | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants.
Statistical Analysis 1: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.6815, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.52 to 1.54]

16. Secondary Outcome: Percentage of Participants With an Event of >/=15% Absolute Decrease in Percentage of Predicted DLco or Death From Any Cause
Description: DLco (in mL/min/mmHg) is a measure of the gas transfer. Predicted DLco is based on sex, age, and height of a person. Percent of predicted DLco (in %) = [(observed DLco)/(predicted DLco)]*100.
Time Frame: Baseline up to the event of >/=15% absolute decrease in percentage of predicted DLco or death from any cause (up to Week 122)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 76 | 76 | 175 | 173
percentage of participants | 9.2 | 6.6 | 14.9 | 11.0

17. Secondary Outcome: Time to First Event of >/=15% Absolute Decrease in Percentage of Predicted DLco or Death From Any Cause
Description: DLco is a measure of the gas transfer. Predicted DLco is based on sex, age, and height of a person. Percent of predicted DLco (in %) = [(observed DLco)/(predicted DLco)]*100. Time from randomization to first occurrence of >/=15% absolute decrease in percentage of predicted DLco or death from any cause was reported. The median time to event was estimated using Kaplan-Meier method. 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 16
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 76 | 76 | 175 | 173
weeks | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to high number of censored participants.
Statistical Analysis 1: Comparison: Monotherapy (Cohort A): Placebo vs Monotherapy (Cohort A): Lebrikizumab; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.5685, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.23 to 2.26]
Statistical Analysis 2: Comparison: Combination Therapy (Cohort B): Placebo + Pirfenidone vs Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone; Stratified Analysis: stratified by baseline FVC (<50%, 50 to 75%, >75%); Test type: Superiority; p = 0.1976, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.37 to 1.23]

18. Secondary Outcome: Percentage of Participants With Anti-therapeutic Antibody (ATA) to Lebrikizumab
Description: ATA to lebrikizumab was tested using a validated immunoassay. A positive ATA result was defined as one in which the presence of detectable ATAs could be confirmed by competitive binding with lebrikizumab. Percentage of participants with positive results for ATA at Baseline and at post-baseline time points were reported. Only participants who received lebrikizumab were included in the analysis.
Time Frame: Baseline and Post-Baseline (assessed at multiple time points: Weeks 4, 12, 24, 36, 52, 56, 64, 76, and at safety follow-up up to Week 122)
Population: Analysis was performed on Safety Population (all participants who received at least one dose of study drug grouped according to the actual treatment received). 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure; 'Number Analyzed' = number of participants evaluable at indicated time points.
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 75 | 172
percentage of participants
  Baseline: number analyzed (Participants) | 75 | 171
  Baseline | 5.3 | 1.8
  Post-Baseline | 6.7 | 5.2

19. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Lebrikizumab at Week 52
Description: Participants who received lebrikizumab were only included in the analysis.
Time Frame: Predose (Hour 0) at Week 52
Population: Analysis was performed on Pharmacokinetic (PK)-Evaluable Population, which included all participants who received at least one dose of study drug and had at least one non-missing PK observation. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure at Week 52.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 62 | 137
micrograms per milliliter (mcg/mL) | 29.6 (14.0) | 25.2 (12.7)

20. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Lebrikizumab
Description: Participants who received lebrikizumab were only included in the analysis.
Time Frame: Predose (Hour 0) at Weeks 4, 12, 24, and 36
Population: Analysis was performed on PK-Evaluable Population. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 78 | 174
mcg/mL
  Cmin at Week 4: number analyzed (Participants) | 74 | 170
  Cmin at Week 4 | 14.0 (4.86) | 14.9 (5.75)
  Cmin at Week 12: number analyzed (Participants) | 68 | 165
  Cmin at Week 12 | 24.4 (9.86) | 25.0 (11.0)
  Cmin at Week 24: number analyzed (Participants) | 65 | 153
  Cmin at Week 24 | 28.5 (12.5) | 25.7 (12.4)
  Cmin at Week 36: number analyzed (Participants) | 61 | 146
  Cmin at Week 36 | 29.9 (14.1) | 25.6 (13.8)

21. Secondary Outcome: Elimination Half-Life (t1/2) of Lebrikizumab
Description: Elimination half-life is the time measured for the plasma drug concentration to decrease by one-half during the elimination phase of the drug. Analysis was performed on PK-Evaluable Population. Participants who received lebrikizumab were only included in the analysis.
Time Frame: Pre-dose (Hour 0) at Weeks 1, 4, 12, 24, 36, 64, 76, 88, 104; and at 4, 12, and 18 weeks post-last dose (last dose = Week 104)
Population: Analysis was performed on PK-Evaluable Population. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
Number analyzed (Participants) | 35 | 125
days | 23.5 (5.36) | 21.9 (4.79)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 122
Description: Safety Population
Arm/Group | Monotherapy (Cohort A): Placebo | Monotherapy (Cohort A): Lebrikizumab | Combination Therapy (Cohort B): Placebo + Pirfenidone | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone
All-Cause Mortality (participants affected / at risk) | 4/76 | 4/78 | 15/177 | 7/174
Serious Adverse Events (participants affected / at risk) | 19/76 | 23/78 | 47/177 | 56/174
Other Adverse Events (participants affected / at risk) | 70/76 | 73/78 | 158/177 | 142/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (Cohort A): Placebo (N=76) | Monotherapy (Cohort A): Lebrikizumab (N=78) | Combination Therapy (Cohort B): Placebo + Pirfenidone (N=177) | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone (N=174)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 3 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0 | 2 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 3 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 4 | 2 | 1
Lung infection (Infections and infestations) | 0 | 1 | 1 | 2
Pneumonia (Infections and infestations) | 2 | 3 | 7 | 7
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 5
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung Adenocarcinoma Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung squamous cell carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 22 | 17
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (Cohort A): Placebo (N=76) | Monotherapy (Cohort A): Lebrikizumab (N=78) | Combination Therapy (Cohort B): Placebo + Pirfenidone (N=177) | Combination Therapy (Cohort B): Lebrikizumab + Pirfenidone (N=174)
Cataract (Eye disorders) | 2 | 4 | 7 | 4
Dry eye (Eye disorders) | 0 | 4 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 2 | 4 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4 | 4 | 6
Constipation (Gastrointestinal disorders) | 11 | 11 | 12 | 14
Diarrhoea (Gastrointestinal disorders) | 16 | 17 | 23 | 18
Dry mouth (Gastrointestinal disorders) | 0 | 6 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 5 | 8
Flatulence (Gastrointestinal disorders) | 0 | 4 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 9 | 9
Nausea (Gastrointestinal disorders) | 10 | 10 | 23 | 28
Toothache (Gastrointestinal disorders) | 4 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 6 | 3 | 9 | 8
Asthenia (General disorders) | 2 | 5 | 3 | 0
Chest discomfort (General disorders) | 5 | 2 | 3 | 3
Chest pain (General disorders) | 5 | 7 | 7 | 10
Fatigue (General disorders) | 12 | 15 | 22 | 28
Injection site erythema (General disorders) | 1 | 4 | 1 | 1
Oedema peripheral (General disorders) | 2 | 4 | 4 | 3
Pain (General disorders) | 2 | 4 | 2 | 1
Bronchitis (Infections and infestations) | 11 | 15 | 11 | 17
Influenza (Infections and infestations) | 4 | 5 | 10 | 3
Lower respiratory tract infection (Infections and infestations) | 5 | 11 | 13 | 10
Nasopharyngitis (Infections and infestations) | 19 | 17 | 25 | 31
Pneumonia (Infections and infestations) | 3 | 1 | 9 | 3
Respiratory tract infection (Infections and infestations) | 5 | 4 | 9 | 8
Rhinitis (Infections and infestations) | 4 | 4 | 7 | 2
Sinusitis (Infections and infestations) | 5 | 6 | 9 | 11
Upper respiratory tract infection (Infections and infestations) | 13 | 18 | 38 | 31
Urinary tract infection (Infections and infestations) | 5 | 9 | 11 | 6
Fall (Injury, poisoning and procedural complications) | 6 | 4 | 3 | 6
Forced vital capacity decreased (Investigations) | 4 | 11 | 6 | 6
Weight decreased (Investigations) | 5 | 2 | 9 | 11
Decreased appetite (Metabolism and nutrition disorders) | 5 | 9 | 22 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 9 | 8 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 12 | 11 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6 | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 5 | 8 | 2
Dizziness (Nervous system disorders) | 10 | 14 | 14 | 11
Headache (Nervous system disorders) | 9 | 10 | 17 | 11
Anxiety (Psychiatric disorders) | 5 | 3 | 1 | 2
Insomnia (Psychiatric disorders) | 3 | 7 | 4 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 21 | 46 | 33
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 18 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 4 | 5
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 10 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 5 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 8 | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 6 | 3 | 24 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 12 | 8
Rash (Skin and subcutaneous tissue disorders) | 5 | 9 | 21 | 18
Hypertension (Vascular disorders) | 4 | 4 | 4 | 7
Pyrexia (General disorders) | 2 | 6 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT01872689/Prot_SAP_000.pdf